CLINICAL TRIAL: NCT02338310
Title: Trial of Perioperative Endocrine Therapy - Individualising Care
Acronym: POETIC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2007/10015; 2007-003877-21 (EudraCT Number); CRUK/07/015 (Other Grant/Funding Number: Cancer Research UK); 08/H1102/37 (Other: Main Research Ethics Committee Number); 63882543 (Registry Identifier: ISRCTN); CCR 2973 (Other: Sponsor)
Record Dates: First submitted 2014-09-16; First posted 2015-01-14 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Anastrozole; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Aromatase Inhibitor (No Intervention): No aromatase inhibitor given around the time of surgery
- Aromatase Inhibitor (Experimental): Aromatase Inhibitor given perioperatively for 4 weeks (two weeks before and two weeks after surgery) Choice of AI is according to centre policy and may be either anastrozole (1mg/day) or letrozole (2.5mg/day)
  Interventions: Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Aromatase Inhibitors — Choice of AI is according to centre policy; any brand can be used
  Other Names: Anastrazole; Letrozole
  Arms: Aromatase Inhibitor

SUMMARY:
To determine whether perioperative endocrine therapy with an aromatase inhibitor (AI) followed by standard adjuvant therapy improves outcome compared with standard adjuvant therapy alone in postmenopausal women with hormone receptor positive breast cancer.

To determine whether the proliferation marker Ki67 as measured by immunohistochemistry (IHC) in the excised cancer around 2 weeks after starting AI therapy will predict for time to recurrence (TTR) in the individual patient more effectively than the pre-treatment Ki67 value.

To determine whether molecular profiling 2 weeks after starting endocrine therapy predicts for long-term outcome in postmenopausal women with hormone receptor positive breast cancer better than at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Post menopausal women with core biopsy-proven hormone receptor positive invasive breast cancer. Postmenopausal is defined as a woman aged ≥50 years fulfilling any one of the following criteria:

   i) with amenorrhoea >12 months and an intact uterus; ii) has undergone a bilateral oophorectomy; iii) in women who have undergone a hysterectomy, then FSH levels within the postmenopausal range (utilising ranges from the testing laboratory facility) are required if the patient is aged <55 years; or iv) in women who have been on HRT within the last 12 months and therefore not amenorrhoeic, FSH levels within the postmenopausal range (utilising ranges from the testing laboratory facility) are required if the patient is aged <55 years.
2. No evidence of metastatic spread by standard assessment according to local guidelines
3. Standard adjuvant endocrine therapy indicated
4. A palpable tumour of any size , or a tumour with an ultrasound size of at least 1.5cm
5. WHO performance status of 0 or 1
6. Written informed consent to participate in the trial and to donation of tissue (fresh tissue and surplus tissue from diagnostic procedures) and blood samples.

Exclusion Criteria:

1. Locally advanced/inoperable breast cancer
2. Evidence of metastatic disease
3. Previous invasive breast cancer (surgically treated DCIS or LCIS allowed)
4. Current bilateral breast cancer
5. Multiple unilateral tumours with different ER/PgR/HER2 status, grade or type (e.g. ductal vs lobular) i.e. anything that suggests two or more different cancers. Multifocal disease with homogenous ER/PgR/HER2 status, grade and type is allowed if at least one lesion is palpable or at least 1.5cm on ultrasound; the largest lesion should be used for sample collection and CRF completion.
6. Concurrent use (defined as use within 4 weeks prior to diagnostic tissue sample being taken) of HRT or any other oestrogen-containing medication (including vaginal oestrogens)
7. Previous use of oestrogen implants at ANY time
8. Prior endocrine therapy or chemotherapy for breast cancer
9. Any invasive malignancy diagnosed within previous 5 years (other than basal cell carcinoma or cervical carcinoma in situ)
10. Any severe co-incident medical disease, inability to give informed consent or unavailability for follow-up
11. Treatment with an unlicensed or investigational drug within 4 weeks before randomisation
12. Current, continuous, long term systemic steroid usage

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4486 (Actual)
Dates: Start 2008-09; Primary Completion 2024-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Time to recurrence | 5 years post-randomisation
  Time to recurrence (TTR) is defined as time from randomisation to local, regional, or distant tumour recurrence or death from breast cancer without prior notification of relapse. Second primary cancers and intercurrent deaths will be treated as censoring events. Patients who are alive and disease free will be censored at the date last seen alive.

SECONDARY OUTCOMES:
Relapse free survival | 5 years post-randomisation
  Second primary cancers and deaths from non-breast cancer causes in the absence of breast cancer relapse will be treated as censoring events.
Time to local recurrence | 5 years post-randomisation
Time to distant recurrence | 5 years post-randomisation
Overall Survival | 5 years post-randomisation
Breast cancer free survival | 5 years post-randomisation
Proliferation rate (Ki67) | At time of surgery (around 2 weeks post-randomisation)
  Comparison of the predictive value of Ki67 at surgery in the perioperative therapy and non perioperative therapy groups will be undertaken using Cox regression, comparing the estimates of the hazard ratios obtained in each treatment group.
Gene expression profile | At time of surgery (around 2 weeks post-randomisation)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Smith, Professor, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (128):
- United Kingdom (128):
  - Ulster Hospital, Dundonald, Belfast
  - Heatherwood and Wexham Park Hospitals NHS trust, Slough, Berkshire
  - Stoke Mandeville Hospital, Aylesbury, Buckinghamshire
  - Prince Philip Hospital, Llanelli, Carmarthenshire
  - Craigavon Area Hospital, Portadown, Co.Amagh
  - Wansbeck General Hospital, Ashington, England
  - North Devon District Hospital, Barnstaple, England
  - City Hospital - Birmingham, Birmingham, England
  - Royal Blackburn Hospital, Blackburn, England
  - Pilgrim Hospital, Boston, England
  - Bradford Teaching Hospitals NHS Trust, St Luke's Hospital, Bradford, England
  - Burnley General Hospital, Burnley, England
  - Cumberland Infirmary, Carlisle, England
  - Chelmsford and Essex Centre, Chelmsford, England
  - Countess of Chester Hospital, Chester, England
  - Chesterfield Royal Hospital, Chesterfield, England
  - Essex County Hospital, Colchester, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Russells Hall Hospital, Dudley, England
  - Wycombe General Hospital, High Wycombe, England
  - Airedale General Hospital, Keighley, England
  - Kidderminster Hospital, Kidderminster, England
  - Whittington Hospital, London, England
  - Royal Free Hospital, London, England
  - Guy's Hospital, London, England
  - King's College Hospital, London, England
  - Royal Marsden - London, London, England
  - St. Mary's Hospital, London, England
  - Wythenshawe Hospital, Manchester, England
  - North Manchester General Hospital - Penine Actute Hospitals Trust, Manchester, England
  - North Tyneside Hospital, North Shields, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - George Eliot Hospital, Nuneaton, England
  - Royal Oldham Hospital, Oldham, England
  - Poole Hospital, Poole Dorset, England
  - Royal Berkshire Hospital, Reading, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Royal Marsden Hosital,, Sutton, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - Royal Hampshire County Hospital, Winchester, England
  - New Cross Hospital, Wolverhampton, England
  - Worcester Royal Hospital, Worcester, England
  - Yeovil District Hospital, Yeovil, England
  - St Margaret's Hospital, Epping, Essex
  - Cheltenham General Hospital, Gloucester, Gloucs
  - St Albans City Hospital, St Albans, Hertfordshire
  - Queen Elizabeth II Hospital, Welwyn Garden City, Hertfordshire
  - Medway Maritime Hospital, Gillingham, Kent
  - Princess Royal University Hospital, Orpington, Kent
  - Tunbridge Wells Hospital, Royal Tunbridge Wells, Kent
  - Grantham and District Hospital, Grantham, Lincolnshire
  - University Hospital, Lewisham, Lewisham, London
  - Queen Elizabeth Hospital, Woolwich, London
  - Ealing Hospital, Southall, Middlesex
  - Royal Victoria Infirmary, Newcastle, Newcastle-Upon-Tyne
  - Harrogate District Hospital, Harrogate, North Yorkshire
  - Belfast City Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Dumfries & Galloway Royal Infirmary, Dumfries, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Princess Royal Hospital, Telford, Shropshire
  - Weston General Hospital, Avon, Weston-super-Mare, Somerset
  - Barnsley District General Hospital, Barnsley, South Yorkshire
  - Rotherham District General Hospital, Rotherham, South Yorkshire
  - Ashford and St Peter's Hospitals, Chertsey, Surrey
  - Kingston Hospital, Kingston upon Thames, Surrey
  - East Surrey Hospital, Redhill, Surrey
  - Bronglais District General Hospital, Aberystwyth, Wales
  - Withybush General Hospital, Haverfordwest, Wales
  - North Wales CTC, Glan Clwyd Hospital, Rhyl, Wales
  - Singleton Hospital, Swansea, Wales
  - Neath Port Talbot Hospital, Port Talbot, West Glamorgan
  - Tameside General Hospital, Ashton-under-Lyne
  - Ysbyty Gwynedd, Bangor
  - Royal United Hospital, Bath
  - Queen Elizabeth Hospital, Birmingham
  - Royal Bolton Hospital, Bolton
  - Royal Bournemouth General Hospital, Bournemouth
  - Bristol Royal Infirmary, Bristol
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - East Kent Hospitals, Canterbury
  - University Hospital Of Wales, Cardiff
  - Castle Hill Hospital, Cottingham
  - University Hospital Coventry, Coventry
  - Leighton Hospital, Crewe
  - Darent Valley Hospital, Dartford
  - Royal Derby Hospital, Derby
  - Royal Devon and Exeter Hospital, Exeter
  - Frimley Park Hospital, Frimley
  - Western Infirmary, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Hereford County Hospital, Hereford
  - Huddersfield Royal Infirmary, Huddersfield
  - Ipswich Hospital, Ipswich
  - Leeds General Infirmary/ St James' University Hospital, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Lincoln County Hospital, Lincoln
  - Royal Liverpool University Hospital, Liverpool
  - Homerton University Hospital, London
  - Charing Cross Hospital, London
  - Northwick Park Hospital, London
  - St Bartholomew's Hospital, London
  - Luton and Dunstable Hospital, Luton
  - Macclesfield District General Hospital, Macclesfield
  - Maidstone Hospital, Maidstone
  - Hillingdon Hospital, Middlesex
  - Milton Keynes General Hospital, Milton Keynes
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Derriford Hospital, Plymouth
  - Dorset County Hospital, Poole
  - Queen's Hospital,, Romford
  - Salford Royal Hospital, Salford
  - Salisbury District Hospital, Salisbury
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Staffordshire General Hospital, Stafford
  - Stepping Hill Hospital, Stockport
  - University Hospital of North Tees, Stockton-on-Tees
  - Musgrove Park Hospital, Taunton
  - St George's Hospital,, Tooting
  - Torbay District General Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Mid Yorkshire Hospitals, Wakefield
  - Warwick Hospital, Warwick
  - Royal Albert Edward Infirmary, Wigan
  - Worthing Hospital, Worthing

REFERENCES:
- [Derived] Smith I, Robertson J, Kilburn L, Wilcox M, Evans A, Holcombe C, Horgan K, Kirwan C, Mallon E, Sibbering M, Skene A, Vidya R, Cheang M, Banerji J, Morden J, Sidhu K, Dodson A, Bliss JM, Dowsett M. Long-term outcome and prognostic value of Ki67 after perioperative endocrine therapy in postmenopausal women with hormone-sensitive early breast cancer (POETIC): an open-label, multicentre, parallel-group, randomised, phase 3 trial. Lancet Oncol. 2020 Nov;21(11):1443-1454. doi: 10.1016/S1470-2045(20)30458-7. PMID 33152284